CLINICAL TRIAL: NCT01165775
Title: Continuous Glucose Monitoring in Pregnant Women Undergoing Betamethasone Therapy
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Professor, Stanford University
Other Study IDs: SU-07082010-6490; 18962 (Other: Stanford University IRB)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Threatened pre term labor patients: Patients receiving betamethasone to minimize the complications of prematurity will monitor blood glucose levels using the Dexcom Seven Plus Continuous Glucose Monitoring System.
  Interventions: Device: Dexcom Seven Plus Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Dexcom Seven Plus Continuous Glucose Monitoring System — Soft sensor for continuous glucose monitoring inserted for up to 24 hours prior to administration of betamethasone. Device to be worn for duration of hospitalization or up to 7 days total, whichever time period is shorter.

SUMMARY:
We hope to clarify how betamethasone affects glucose levels in the mother in the days after receiving the drug. This understanding will hopefully allow us to better anticipate the risk of maternal hyperglycemia and therefore establish more appropriate monitoring of maternal glucose to prevent maternal and neonatal complications of hyperglycemia.

DETAILED DESCRIPTION:
Pregnant patients who are undergoing inpatient betamethasone therapy as part of their clinical care will be eligible for the study. Once the clinical team and patients have agreed to pursue betamethasone therapy, the patients' treating physician or nurse will inquire if the patient is interested in participating in our study protocol. Those patients who are interested in participation will be consented by either a member of the treatment team or the study team. Prior to receiving the first betamethasone dose, a soft sensor for continuous glucose monitoring system (CGMS) will be inserted superficially under the skin. For those patients who will be receiving a scheduled course of betamethasone, the sensor may be inserted up to 24 hours prior to the betamethasone administration. The patient will be instructed on how to wear and care for the device. She will wear the CGMS for the duration of her hospitalization or for up to 7 days total, whichever time period is shorter. For those patients who are diabetic, they will receive normal finger stick blood glucose (FSBG) monitoring and insulin therapy as determined by their treating physicians. Those patients who are not diabetic will need to have 2 FSBG checks each day to correlate with the device. Abnormal values will be reported to the patients' treating physician and addressed by the treating physician. Prior to being discharged from the hospital, the patient will have the device removed. The patient will otherwise be treated routinely. We will record baseline demographic information and medical history from each of the women. We will also record information from the neonates' newborn medical records.

ELIGIBILITY:
Inclusion Criteria:- 18 years of age or older

* Receiving betamethasone as part of routine clinical care.
* Pregnancy between 23+5 and 35+0 weeks Exclusion Criteria:- Less than 18 years old.
* Major fetal anomalies
* Use of steroid medications in the past 2 weeks.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women receiving betamethasone
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Langen ES, Kuperstock JL, Sung JF, Taslimi M, Byrne J, El-Sayed YY. Maternal glucose response to betamethasone administration. Am J Perinatol. 2015 Feb;30(2):143-8. doi: 10.1055/s-0034-1376387. Epub 2014 Jun 10. PMID 24915559
- See also: Maternal glucose response to betamethasone administration — http://dx.doi.org/10.1016/j.ajog.2011.10.211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women receiving clinically indicated betamethasone between 24 and 34 weeks of pregnancy were recruited from the labor and delivery setting.
Period: Overall Study
Arm/Group | Threatened Pre Term Labor Patients
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Women receiving clinically indicated betamethasone between 24 and 34 weeks of pregnancy. Data are available for 15 of 17 participants.
Groups:
- Threatened Pre Term Labor Patients: Patients receiving betamethasone to minimize the complications of prematurity will monitor blood glucose levels using the Dexcom Seven Plus Continuous Glucose Monitoring System.
  Dexcom Seven Plus Continuous Glucose Monitoring System: Soft sensor for continuous glucose monitoring inserted for up to 24 hours prior to administration of betamethasone. Device to be worn for duration of hospitalization or up to 7 days total, whichever time period is shorter.
  Data are available for 15 of 17 participants.
Arm/Group | Threatened Pre Term Labor Patients
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Gestational age at enrollment [Mean (Full Range); unit: weeks] | 29.29 [25.14 to 34.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage Time Spent Above Glucose Thresholds (>110;>144;>180) 24-48 Hours Post Betamethasone Treatment
Description: During a 24 hour monitoring period (24-48 hours post betamethasone treatment), which percentage of the time was spent above glucose thresholds (>110;>144;>180)
Time Frame: 24-48 hours post betamethasone treatment
Population: Seventeen women were enrolled at the time of betamethasone administration and data were available for 15 patients.
Measure: Mean (Standard Deviation); unit: percentage time
Groups:
- Non-Diabetic Threatened Pre Term Labor Patients; Diabetic Threatened Pre Term Labor Patients: Patients receiving betamethasone to minimize the complications of prematurity will monitor blood glucose levels using the Dexcom Seven Plus Continuous Glucose Monitoring System.
  Dexcom Seven Plus Continuous Glucose Monitoring System: Soft sensor for continuous glucose monitoring inserted for up to 24 hours prior to administration of betamethasone. Device to be worn for duration of hospitalization or up to 7 days total, whichever time period is shorter.
Arm/Group | Non-Diabetic Threatened Pre Term Labor Patients | Diabetic Threatened Pre Term Labor Patients
Number analyzed (Participants) | 11 | 4
percentage time
  mean (SD)% time with blood glucose > 110 | 73 (6) | 79 (20)
  mean (SD)% time with blood glucose > 144 | 40 (17) | 58 (26)
  mean (SD)% time with blood glucose > 180 | 17 (13) | 24 (13)

2. Secondary Outcome: Neonatal Hypoglycemia
Time Frame: birth to discharge
Population: Neonates from birth to discharge. The maternal patients received betamethasone to minimize the complications of prematurity. Maternal blood glucose levels were monitored using the Dexcom Seven Plus Continuous Glucose Monitoring System.
Measure: Number; unit: participants
Groups:
- Neonates With Hypoglycemia: Neonates with hypoglycemia from birth to hospital discharge.
- Neonates Without Hypoglycemia: Neonates without hypoglycemia from birth to hospital discharge.
- Neonates With Unknown Hypoglycemia Status: Neonates with unknown hypoglycemia status from birth to hospital discharge.
Arm/Group | Neonates With Hypoglycemia | Neonates Without Hypoglycemia | Neonates With Unknown Hypoglycemia Status
Number analyzed (Participants) | 4 | 6 | 5
participants
  Maternal Diabetes | 2 | 2 | 0
  No Maternal Diabetes | 2 | 4 | 5
Statistical Analysis 1: Comparison: Neonates With Hypoglycemia vs Neonates Without Hypoglycemia vs Neonates With Unknown Hypoglycemia Status; Test type: Superiority or Other; p = 0.2155, Chi-squared

ADVERSE EVENTS:
Arm/Group | Threatened Pre Term Labor Patients
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No